CLINICAL TRIAL: NCT05695833
Title: Comparative Study Between Long Pulsed Nd:YAG Laser and Radiofrequency in Treatment of Fingernail Psoriasis
Brief Title: Nd:YAG Laser and Radiofrequency in Treatment of Fingernail Psoriasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar El Sayed, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Radiofrequency nail psoriasis
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Nail Psoriasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency (Experimental): Device
  Interventions: Device: Radiofrequency
- Nd Yag Laser (Active Comparator): Device
  Interventions: Device: Radiofrequency

INTERVENTIONS:
Device: Radiofrequency — Device emitting electric waves generating heat

SUMMARY:
Compare the effect of Radiofrequency to long pulsed Nd:YAG 1064 nm laser in treatment of fingernail psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Nail Psoriasis

Exclusion Criteria:

* Manual workers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-20 (Estimated); Primary Completion 2023-04-20 (Estimated); Study Completion 2023-05-20 (Estimated)

PRIMARY OUTCOMES:
Targeted Nail Psoriasis Severity Index (tNAPSI) score | 12 weeks

REFERENCES:
- [Derived] El-Basiony MAS, El-Komy MHM, Samy NA, Aly DG, El-Gendy H, Soliman MM, Abdel Salam Hassan MF, El Sayed H. Efficacy of Nonablative Bipolar Radiofrequency in the Treatment of Fingernail Psoriasis. Dermatol Surg. 2025 May 1;51(5):522-526. doi: 10.1097/DSS.0000000000004531. Epub 2024 Dec 16. PMID 39679566